CLINICAL TRIAL: NCT05947799
Title: A Comparative Study on the Effectiveness of Video vs Text-Based Education in Heart Failure
Acronym: EDUCATE-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alexander Sandhu, Instructor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69691
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure
Keywords: Heart Failure Education
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Video medication module then text self-monitoring module (Other): Patients are provided education via an online animated video on heart failure medications followed by a online text document on heart failure self-monitoring.
  Interventions: Other: Baseline questionnaires; Other: Post-questionnaire
- Text medication module then video self-monitoring module (Other): Patients are provided education via an online text document on heart failure medications followed by a online animated video on heart failure self-monitoring.
  Interventions: Other: Baseline questionnaires; Other: Post-questionnaire
- Video self-monitoring module then text medication module (Other): Patients are provided education via an online animated video on heart failure self-monitoring followed by a online text document on heart failure medications.
  Interventions: Other: Baseline questionnaires; Other: Post-questionnaire
- Text self-monitoring module then video medication module (Other): Patients are provided education via an online text document on heart failure self-monitoring followed by a online animated video on heart failure medication management.
  Interventions: Other: Baseline questionnaires; Other: Post-questionnaire

INTERVENTIONS:
Other: Baseline questionnaires — Questionnaires asking about the participant's familiarity with heart failure medication and management before watching/reading the educational modules.
Other: Post-questionnaire — Questionnaires asking about the participant's familiarity with heart failure medication and management after watching/reading the educational modules.

SUMMARY:
This is a study seeking to compare the change in overall heart failure (HF) knowledge score and participant preference between video-based and text-based HF education modules. Participants will be randomized to watching and reading different combinations of video-based education modules and text-based education modules. Participants will be asked to answer questions about their familiarity with heart failure medications and management before and after the said education modules.

DETAILED DESCRIPTION:
This study compares the change in heart failure (HF) knowledge and participant preference between video-based and text-based HF education modules. Educational material regarding two different topics - heart failure self-monitoring and medication management - has been developed in two different formats: animated educational videos and text-based documents. Both formats contain the same information. In this study, participants will be randomized to either watching or reading different combinations of the education for these two topics to better understand which educational tool - animated videos or text-based - is preferred by participants and leads to greater educational attainment. Educational attainment is evaluated by pre and post questions about both topics.

ELIGIBILITY:
Inclusion Criteria:

* Participants with heart failure with reduced ejection fraction (EF <50%)

Exclusion Criteria:

* Participants who have the inability to independently read or answer written questions in English and are non-conversant in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Heart Failure Knowledge Score Improvement | Collected immediately following patient educational module completion
  Change in percentage of correct answers on a questionnaire about heart failure knowledge regarding medications and self-management
Patient preference for heart failure education module | Collected immediately following patient educational module completion
  Likert scale of preference between video and text based modules

SECONDARY OUTCOMES:
Change in HF medication score on knowledge assessment between video-based and text-based education modules | Collected immediately following patient educational module completion
  Change in percentage of correct answers on a questionnaire related to heart failure medications
Change in HF self-management score on knowledge assessment between video-based and text-based education modules | Collected immediately following patient educational module completion
  Change in percentage of correct answers on a questionnaire related to heart failure self-management
Change in self-assessed knowledge of HF medications between video-based and text-based education modules | Collected immediately following patient educational module completion
  Difference in Likert scale of self-assessed knowledge of HF medications before and after educational modules
Change in self-assessed knowledge of HF self-monitoring between video-based and text-based education modules | Collected immediately following patient educational module completion
  Difference in Likert scale of self-assessed knowledge of HF self-monitoring before and after educational modules

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Sandhu, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital & Clinics, Stanford, California, United States